CLINICAL TRIAL: NCT00737633
Title: An Open-Label, Non-Randomized Multicenter Study to Evaluate the Long-Term Safety and Efficacy of VI-0521 in Providing and Maintaining Glycemic Control in Type 2 Diabetic Adults
Brief Title: Open-Label Study to Evaluate the Long-Term Safety and Efficacy of VI-0521 in Type 2 Diabetic Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited regulatory value to uncontrolled trials. No safety/efficacy concerns.
Sponsor: VIVUS LLC (Industry)
Collaborators: Synteract, Inc. (Industry); Sentrx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM-231
Record Dates: First submitted 2008-08-17; First posted 2008-08-19 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes
Keywords: Diabetes; Type 2 Diabetes; Diabetes Mellitus; Metabolic Diseases; Glucose Metabolism Disorders; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Metabolic Diseases; Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 16-Week population (Experimental): Placebo subjects in OB-202 (NCT00486291) and DM-230 (NCT00600067)
  Interventions: Drug: VI-0521
- 72-Week population (Experimental): Active treatment subjects in OB-202 (NCT00486291) and DM-230 (NCT00600067)
  Interventions: Drug: VI-0521

INTERVENTIONS:
Drug: VI-0521 — Phentermine 15 mg/Topiramate controlled release (CR) 92 mg, oral capsule, once daily, 58 weeks

SUMMARY:
This study is an extension of a study that has been ongoing for 1 year. The purpose of this open label study is to see the how well type 2 diabetics respond to VI-0521(phentermine/topiramate) in controlling blood sugar and how safe VI-0521 is over an extended period of time. All subjects eligible to enroll into this study will receive study drug.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the qualifying DM-230 trial
* If females of child-bearing potential, subjects must be using adequate contraception
* Provide written informed consent
* Be willing and able to comply with scheduled study visits, treatment plan, lab tests and other study procedures
* Be greater than 80% compliant in study medication use during the last three visits for DM-230

Exclusion Criteria:

* Subjects who have developed one or more morbidities during the DM-230 trial that would pose a safety concern

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Troupin, MD, MBA, Study Director — VIVUS LLC
Locations (9):
- United States (9):
  - Research Site, Birmingham, Alabama
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Spring Valley, California
  - Research Site, Walnut Creek, California
  - Research Site, Bethesda, Maryland
  - Research Site, Austin, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an extension study to OB-202 (NCT00486291) and DM-230 (NCT00600067)
Period: Overall Study
Arm/Group | 16-week Population | 72-week Population
Started | 44 | 57
Completed | 0 | 0
Not Completed | 44 | 57
Not completed — Study terminated by sponsor | 44 | 55
Not completed — Lost to Follow-up | 0 | 1
Not completed — protocol non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 16-week Population: subjects who were randomized to placebo in previous study
- 72-week Population: subjects who were randomized to active during previous study
- Total: Total of all reporting groups
Arm/Group | 16-week Population | 72-week Population | Total
Number analyzed (Participants) | 44 | 57 | 101
Age Continuous [Mean (Standard Deviation); unit: years] | 50.2 (8.6) | 49.5 (7.0) | 49.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 48 | 73
  Male | 19 | 9 | 28
Region of Enrollment [Number; unit: participants]
  United States | 44 | 57 | 101

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 72
Time Frame: Baseline to 72 weeks
Population: Intent-to-treat (ITT)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 16-week Population | 72-week Population
Number analyzed (Participants) | 44 | 57
percent change | -0.5 (0.79) | -1.4 (1.34)

2. Secondary Outcome: Percent Weight Change From Baseline to Week 72
Time Frame: Baseline to 72 weeks
Population: Intent-to-treat (ITT)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 16-week Population | 72-week Population
Number analyzed (Participants) | 44 | 57
percent change | -5.7 (4.64) | -10.1 (8.7)

ADVERSE EVENTS:
Time Frame: AEs were collected from when written informed consent was provided through 28 days after the last dose of investigational product.
Arm/Group | 16-week Population | 72-week Population
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/57
Other Adverse Events (participants affected / at risk) | 33/44 | 34/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 16-week Population (N=44) | 72-week Population (N=57)
Coronary Artery Disease (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 16-week Population (N=44) | 72-week Population (N=57)
upper respiratory tract infection (Infections and infestations) | 3 | 2
gastroenteritis (Infections and infestations) | 2 | 2
sinusitis (Infections and infestations) | 2 | 2
nasopharyngitis (Infections and infestations) | 0 | 3
influenza (Infections and infestations) | 1 | 2
parasthesia (Nervous system disorders) | 2 | 3
dizziness (Nervous system disorders) | 7 | 0
headache (Nervous system disorders) | 3 | 1
dysgeusia (Nervous system disorders) | 6 | 0
nausea (Gastrointestinal disorders) | 4 | 3
diarrhea (Gastrointestinal disorders) | 1 | 3
constipation (Gastrointestinal disorders) | 7 | 0
gastritis (Gastrointestinal disorders) | 0 | 2
dyspepsia (Gastrointestinal disorders) | 1 | 2
dry mouth (Gastrointestinal disorders) | 5 | 1
abdominal distension (Gastrointestinal disorders) | 2 | 1
hypoglycemia (Metabolism and nutrition disorders) | 6 | 8
insomnia (Psychiatric disorders) | 6 | 2
anxiety (Psychiatric disorders) | 2 | 2
fatigue (General disorders) | 6 | 1
irritability (General disorders) | 2 | 1
back injury (Injury, poisoning and procedural complications) | 2 | 0
eye pain (Eye disorders) | 2 | 1
lacrimation increased (Eye disorders) | 2 | 0
chromatopsia (Eye disorders) | 2 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.